#### **INFORMED CONSENT FORM – MOTHER**

Title: Effect of Enhanced Recovery After Cesarean (ERAS) Protocol on Mother-Infant and

Father-Infant Bonding: A Multicenter Randomized Controlled Trial

**Protocol Code:** ERAS-CS-BOND-1

Principal Investigator: Dr. Gökçenur Karakelleoğlu

**Institution:** Istanbul Okan University Hospital

Country: Türkiye

Version: 1.0

Date: November 04, 2025

NCT Number: Not yet Assigned

#### INFORMED CONSENT FORM – MOTHER

Study Title: Effect of Enhanced Recovery After Cesarean (ERAS) Protocol on Mother—

Infant and Father-Infant Bonding

Principal Investigator: Dr. Gökçenur Karakelleoğlu

**Institution:** Istanbul Okan University Hospital

## 1. Purpose of the Study

This study aims to evaluate whether the ERAS protocol improves mother–infant and father–infant bonding after cesarean delivery compared with standard care.

### 2. Study Procedure

After your cesarean birth, you will be randomly assigned to the ERAS group or the standard care group.

At 2 hours, 24 hours, day 4, and day 7 postpartum, you will be asked to complete validated questionnaires (MIBS, PBQ, EPDS).

No medical procedures will be performed as part of the study.

#### 3. Risks/Discomfort

No physical risks exist. Emotional discomfort may occur while answering questionnaires; you may stop at any time.

## 4. Benefits

There may be no direct benefit to you. Findings may improve postpartum care for future mothers.

# 5. Confidentiality

All information will be coded and kept confidential. Your name will not appear in any report. Data stored securely for 15 years.

# 6. Voluntary Participation

Participation is voluntary. You may withdraw at any time without affecting your care.

### 7. Contact

Dr. Gökçenur Karakelleoğlu

Email: gokcenur82@hotmail.com

## **Consent Statement**

"I have read this form. I voluntarily agree to participate."

Mother's Name / Signature / Date

Researcher's Name / Signature / Date